CLINICAL TRIAL: NCT02469883
Title: A Phase I Study of Sinotecean on Tolerance and Pharmacokinetics
Brief Title: A Study of Sinotecean on Tolerance and Pharmacokinetics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XNTK-I-03
Record Dates: First submitted 2015-03-22; First posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sinotecean (Experimental)
  Interventions: Drug: Sinotecean

INTERVENTIONS:
Drug: Sinotecean

SUMMARY:
This study is conducted to assess the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT), to evaluate the pharmacokinetics, safety and preliminary anti-tumor activity of Sinotecean.

ELIGIBILITY:
Inclusion Criteria:

* late malignant tumor patients diagnosed with the pathological and/or cytological;
* lack of the standard treatment or treatment failure;
* 18-65years, ECOG:0-1,expected survival period >3 months;
* main organs function is normal;
* signed and dated informed consent

Exclusion Criteria:

* participated in other clinical trials in four weeks;
* currently under other effective treatment;
* end of anti-tumor treatment within 4 weeks(end of Nitrosourea/Mitomycin within 6 weeks);
* AE ≥ Grade 2(according to NCI-CTC 4.0),except hair loss;
* with ischemic heart disease, heart failure, severe arrhythmia, cerebrovascular disease, asthma, severe infections, active peptic ulcer;
* urine protein: ++, and urinary in 24 hours > 1.0g;
* uncontrolled primary or metastatic brain;
* have immunodeficiency history;
* according to the researcher's judgment,there are concomitant diseases which will seriously endanger the patients or obstruct the patients to complete the clinical trial;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Assessments for Area Under Curve（AUC） | Day 1-2 Single Dose
  To collect point with single drug:5 min/10 min/15 min/30 min/1 h/2h/4h/6 h/8h/10h/12 h/24 h/32h/48 h
Pharmacokinetic Assessments for Cmax | Day 1-2 Single Dose
Pharmacokinetic Assessments for Tmax | Day 1-2 Single Dose

SECONDARY OUTCOMES:
Objective Response Rate （ORR) | each 42 days up to intolerance the toxicity or progression of disease（PD） (up to 24 months)
Maximum tolerated dose(MTD) | up to 24 months
Dose-limiting toxicity(DLT) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China